CLINICAL TRIAL: NCT04058691
Title: Prospective/Retrospective Multicenter Registry to Examine the Real-world Performance in France of the E-vita OPEN PLUS Stent Graft System
Brief Title: Prospective/Retrospective Registry of the E-vita OPEN PLUS Stent Graft System in France
Acronym: FEOR
Status: Completed | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: FEOR
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Vascular Diseases
Keywords: Aortic aneurysms; aortic dissections; thoracic
MeSH Terms: conditions — Vascular Diseases; Aortic Aneurysm; Aortic Dissection | interventions — Sutureless Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Surgical repair — Open surgery
  Other Names: Frozen Elephant Trunk Technique

SUMMARY:
The FEOR registry is undertaken to examine the real-world data of patients that were treated with the E-vita OPEN Plus Stent Graft System under routine care in France. This registry is a requirement of the Haute Autorité de Santé (HAS).

DETAILED DESCRIPTION:
Data Collection on patients who have been implanted with an E-vita OPEN PLUS Stent Graft System from 15th July 2014 until 31st May 2019. The E-vita OPEN PLUS Stent Graft System was implanted at the discretion of the treating physician. Participating physicians provided their observations collected during routine care for patients he/she had decided to treat with the E-vita OPEN PLUS Stent Graft System.

The period of data collection was three years starting from the intervention of each patient. Data verification was performed.

ELIGIBILITY:
Inclusion Criteria:

None

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients with aortic pathologies who have undergone implantation of the E-vita OPEN PLUS Stent Graft System at their physician's discretion since July 15th, 2014.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | 30 days
  The primary endpoint is a composite endpoint of morbi-mortality defined as following:
  * Mortality rate
  * Morbidity rate including neurological complications, visceral malperfusion, and renal complications.
  Neurological complications comprise new cerebrovascular accident (CVA)/stroke, spinal cord ischemia, paraparesis, paraplegia as reported in the eCRF.
  Visceral malperfusion includes new bowel obstruction and visceral ischemia/infarction as reported in the eCRF.
  Renal complications comprise new renal insufficiency and renal insufficiency requiring dialysis as reported in the eCRF.

SECONDARY OUTCOMES:
Mortality | 1 year
  Mortality rate
Mortality | 3 year
  Mortality rate
Morbidity | 1 year
  Morbidity rate
Morbidity | 3 year
  Morbidity rate
Endoleak type Ib | 1 year
  Rate of endoleak type Ib
Endoleak type Ib | 3 year
  Rate of endoleak type Ib
Endoleak type II | 1 year
  Rate of endoleak type II
Endoleak type II | 3 year
  Rate of endoleak type II
Endoleak type III | 1 year
  Rate of endoleak type III
Endoleak type III | 3 year
  Rate of endoleak type III
Endoleak type IV | 1 year
  Rate of endoleak type IV
Endoleak type IV | 3 year
  Rate of endoleak type IV
Adverse Events | 1 year
  Rate of adverse events
Adverse Events | 3 year
  Rate of adverse events
Reinterventions | 1 year
  Rate of reinterventions
Reinterventions | 3 year
  Rate of reinterventions
Secondary interventions | 1 year
  Rate of secondary interventions:
  TAA: A planned additional endovascular intervention with a TAA stent graft in the downstream aorta.
  Treatment of the dissection distally to the targeted pathology that was initially treated using the Evita OPEN PLUS Stent Graft is not a reintervention but an additional intervention (secondary intervention (s)).
Secondary interventions | 3 year
  Rate of secondary interventions:
  TAA: A planned additional endovascular intervention with a TAA stent graft in the downstream aorta.
  Treatment of the dissection distally to the targeted pathology that was initially treated using the Evita OPEN PLUS Stent Graft is not a reintervention but an additional intervention (secondary intervention (s)).
Fully thrombosed false lumen (dissections) | 1 year
  Rate of patients with fully thrombosed false lumen in the stented area (until 2cm proximal from distal end of stent graft)
Fully thrombosed false lumen (dissections) | 3 year
  Rate of patients with fully thrombosed false lumen in the stented area (until 2cm proximal from distal end of stent graft)
Partially thrombosed false lumen (dissections) | 1 year
  Rate of patients with partially thrombosed false lumen in the stented area
Partially thrombosed false lumen (dissections) | 3 year
  Rate of patients with partially thrombosed false lumen in the stented area
Patent false lumen (dissections) | 1 year
  Rate of patients with patent false lumen in the stented area
Patent false lumen (dissections) | 3 year
  Rate of patients with patent false lumen in the stented area

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Verhoye, Prof., Principal Investigator — Rennes Pontchaillou University Medical Centre
Locations (2):
- France (2):
  - Rennes Pontchaillou University Medical Centre, Rennes, Cedex 9
  - Clinique de l'Infirmerie Protestante à Lyon, Caluire-et-Cuire